CLINICAL TRIAL: NCT01944891
Title: Estudo do Estado Nutricional e da Dieta em Raparigas Adolescentes na Zambézia
Brief Title: Diet and Nutritional Status of Adolescent Girls in Zambézia, Mozambique
Acronym: ZANE
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Marja Mutanen, Professor, University of Helsinki
Other Study IDs: 151152
Record Dates: First submitted 2013-08-30; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Nutritional Status; Diet
Keywords: Adolescent girls; Mozambique; Diet; Anthropometrics; Serum biomarkers

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, urine, buccal cells
Oversight: Data Monitoring Committee: No

SUMMARY:
Data on the diet and nutritional status of adolescent girls in Zambézia Province, Mozambique was collected. A cross-sectional study was carried out in 2010 in two seasons, January-February and May-June. Participants (total n=551) were recruited from Quelimane (the provincial capital), Maganja da Costa district and Morrumbala district.

ELIGIBILITY:
Inclusion Criteria:

Girls in the target age range who were able to visit the study centre and didn't have any significant illness preventing participation were considered eligible.

Exclusion Criteria:•

* age not between 15 and 18 years
* any apparent significant illness, disability or unstable medical condition which could lead to difficulty participating in the study
* unwillingness to participate in the study
* unwillingness or inability to arrive at the study location at the requested time.

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent girls living in Quelimane city, Maganja da Costa district and Morrumbala district.
Sampling Method: Probability Sample
Enrollment: 551 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Blood vitamin and mineral concentrations | cross-sectional 2010, single measurement
Dietary assessment | cross-sectional 2010, single measurement
  24-hr recall, food frequency questionnaire

SECONDARY OUTCOMES:
Diseases (intestinal helminths, malaria parasitemia, HIV-status) | cross-sectional 2010, single measurement

CONTACTS AND LOCATIONS:
Overall Officials: Marja L Mutanen, Prof., Principal Investigator — University of Helsinki
Locations (1):
- Department of Food and Environmental Science, University of Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Freese R, Korkalo L, Vessby B, Tengblad S, Vaara EM, Hauta-alus H, Selvester K, Mutanen M. Essential fatty acid intake and serum fatty acid composition among adolescent girls in central Mozambique. Br J Nutr. 2015 Apr 14;113(7):1086-95. doi: 10.1017/S0007114515000306. Epub 2015 Mar 16. PMID 25772191
- [Derived] Korkalo L, Freese R, Fidalgo L, Selvester K, Ismael C, Mutanen M. A Cross-Sectional Study on the Diet and Nutritional Status of Adolescent Girls in Zambezia Province, Mozambique (the ZANE Study): Design, Methods, and Population Characteristics. JMIR Res Protoc. 2014 Mar 5;3(1):e12. doi: 10.2196/resprot.3109. PMID 24598035